CLINICAL TRIAL: NCT00439088
Title: Comparison of the Patient Activity Monitor to a Pedometer During Ambulation Monitoring of Transtibial Amputees
Brief Title: Try Walking a Mile in These Shoes: Activity Level of Lower Extremity Amputees
Acronym: PamPed
Status: Completed | Type: Observational
Sponsor: University of Ottawa (Other)
Other Study IDs: TRC-0020-02
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2007-03

CONDITIONS: Amputee
Keywords: Ambulation; Ambulatory Monitoring; Activities of Daily Living; Pedometer; Validation Studies [PT]

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to compare the accuracies of the Patient Activity Monitor to that of a standard pedometer during a walking task and some day-to-day activities in a simulated apartment setting.

DETAILED DESCRIPTION:
The ability to accurately measure daily activity levels in lower extremity amputee patients is important for a better understanding of their use of prosthetic limbs. Most studies have shown that patients often report their activity level inaccurately. More objective data on activity levels will not only provide information helpful for determining the appropriate prosthetic components for an individual, it will also be helpful when assessing the effects that medical illness have on activity levels and in objectively determining the benefits of rehabilitation. In addition, being able to measure activity accurately will allow further verification of currently developed clinical surveys designed to determine amputee activity in a practical form.

Until more recently a practical, accurate and affordable means of monitoring lower extremity amputee activity has not been available for use. Currently a monitoring device designed specifically for this task is available for research use. It is called the Patient Activity Monitor (PAM). Many different models of more generic activity monitoring devices, called pedometers, also exist and need to be further tested in the amputee population.

The objective of our study was to measure and compare the step count and ambulation distance accuracies of a Yamax Digi-Walker pedometer and the PAM in transtibial amputees at the K3 Level within a simulated apartment setting and during relatively continuous gymnasium walking.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputees who were identified as community level ambulators (K-Level 3)

Exclusion Criteria:

* Malfunction of prosthesis; or
* New medical co-morbidities that impacted on ambulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Meridith B Marks, M.D., M.ed, Study Director — University of Ottawa
Locations (1):
- The Rehabilitation Centre, Ottawa, Ontario, Canada